CLINICAL TRIAL: NCT04350242
Title: Characteristics of Patients With Musculoskeletal Disorders Who Attend a Private Physiotherapy Clinic in Argentina: a Retrospective Study
Brief Title: Characteristics of Patients With Musculoskeletal Disorders
Status: Completed | Type: Observational
Sponsor: Kine Kinesiologia Deportiva y Funcional (Network)
Responsible Party: Principal Investigator, Diego Mendez, Principal Investigator, Physical Therapist., Kine Kinesiologia Deportiva y Funcional
Other Study IDs: 1
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Musculoskeletal Pain; Knee Injuries
MeSH Terms: conditions — Musculoskeletal Pain; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiology, a word derived from the Greek epi (on) demos (people), is a scientific discipline in the area of medicine that studies the distribution, frequency and determining factors of chemical diseases in defined human populations. It is the method of problem solving research used by epidemiologists, scientists, statisticians, doctors, and other health professionals to get to the root of health problems in a community. Beyond the important role of descriptive epidemiology in generating etiological hypotheses, it also provides a description of the frequency and / or patterns of disease occurrence at the individual or social level.

In the field of medicine and physiotherapy, epidemiological studies of musculoskeletal injuries acquire great relevance considering that they are the main cause of disability, increasing their prevalence year after year and carrying high economic and social costs. Worldwide, the Epidemiology of musculoskeletal pathologies has been reported in both the general population and specific populations.

Despite the fact that kinesiology has been an established profession in Argentina since the 1940s, there is an evident lack of scientific information on this discipline. Currently, epidemiological reports of published musculoskeletal pathologies are scarce in our country. To our knowledge, the characteristics of the population of patients with musculoskeletal injuries who attend a private sports kinesiology office are not known. A study of these characteristics could help to better understand this population, improving routine clinical practice, as well as providing a database for the development of future scientific studies.

For this reason, the main objective of this study is to describe the characteristics of the patients who come to an external kinesiology office at a private institution in Argentina. The secondary objective is to evaluate the relationship between the body mass index (BMI) and the affected body regions.

DETAILED DESCRIPTION:
Design Variables related to injury Analytical, cross-sectional and retrospective study will be recorded. Population Those patients who attended a private physiotherapy center in the Autonomous City of Buenos Aires between January 2017 and December 2019 were consecutively included. Those cases in which the affected body region was not recorded were excluded.

Given the characteristics of the study, the signing of the informed consent by the patients was not required.

Process The information used for the analysis was collected during the first session in an evaluation form, prepared by kinesiologists belonging to the institution and used since January 2017. All the professionals who participated in the study had a prior period of theoretical training in the use of the file and the registration of the data. The information of each patient was collected by kinesiologists from this institution and posted on a Microsoft Excel® spreadsheet from which the corresponding analyzes were performed.

Sociodemographic variables The following variables will be recorded: sex, age, weight, height, body mass index (BMI), laterality, main sport, smoking, hours of rest and quality of self-perceived sleep (good, fair or poor).

The following variables: affected body region, type of injury, duration and form of onset of symptoms (acute without apparent reason, acute by specific event, gradual without apparent reason and gradual by specific event).

Statistic analysis Categorical variables are reported as presentation number and percentage. Continuous variables that assume a symmetric distribution are reported as mean ± standard deviation, while those with asymmetric distribution as median and interquartile range (RIC 25-75). A univariate analysis was used to search for the association between BMI and probability of injury. The R Markdown program was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

All patients who attended a private physiotherapy center in the Autonomous City of Buenos Aires, between January 2017 and December 2019.

Criteria Exclusion:

* Cases where the affected body region was not recorded were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of private physiotherapy clinic
Sampling Method: Probability Sample
Enrollment: 1539 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of body region injured | January 2018 - January 2020
  Distribution of affected body region of the population

SECONDARY OUTCOMES:
Age | January 2018 - January 2020
  Mean age of population
Sex | January 2018 - January 2020
  Female or male
Body mass index | January 2018 - January 2020
  Calculation using a person's height and weight

CONTACTS AND LOCATIONS:
Locations (1):
- KINÉ kinesiología deportiva y funcional, CABA, Argentina

IPD SHARING:
Plan to Share IPD: Undecided